CLINICAL TRIAL: NCT06022016
Title: Study of Families With an Hemopathies Predisposition Related to the DDX41 Gene.
Acronym: LUCID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23HEMA06
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: DDX41 Gene Mutation
Keywords: GermlIne DDX41 mutation; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Idiopathic Cytopenia; LeUkemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia | interventions — Association

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Index case or related (Experimental)
  Interventions: Genetic: For each person (index case or related) included in this study:

INTERVENTIONS:
Genetic: For each person (index case or related) included in this study: — * an health questionnaire will be completed in order to gather information on the participant's medical history and lifestyle.
  * a saliva sample will be taken (if applicable) so that a genetic analysis can be performed.

SUMMARY:
This is a multicenter, interventional, historico-prospective cohort pilot study aimed at specifying the phenotype of subjects carrying a constitutional familial DDX41 mutation, with a view to eventually publishing oncogenetic recommendations for carriers of this mutation.

The main objective of the LUCID project is to assess the cumulative risk of hematological diseases as a function of age in DDX41 germline mutation carriers.

This study will be carried out in two stages:

Stage 1: Inclusion of index cases in an oncogenetic consultation (salivary test, completion of an health self-questionnaire and collection of contact details for the related cases).

Stage 2: Proposition of participation to family members, by correspondence, and determination of carrier or non-carrier status of the constitutional familial DDX41 mutation (based on a salivary test).

A maximum of 210 index case patients and 700 family member will be included in this study.

ELIGIBILITY:
Index cases:

Inclusion Criteria:

1. Women or man aged ≥ 18 years old.
2. Personal history(s) of hemopathy or patient with hemopathy at the time of inclusion.
3. Patient with a tumor mutation of DDX41 with an allelic frequency (AF) ≥ 30% (with total depth of nucleotide position >300x: provide tumor molecular analysis report).

   Special case of inclusion of deceased index cases: the DDX41 tumor mutation of interest must be accompanied by another somatic DDX41 mutation (the most frequent being p.R525H).

   Or patient known to be a constitutional carrier of a DDX41 mutation confirmed after oncogenetic consultation (in this case, provide constitutional analysis report).
4. Patient (or beneficiary) agreeing to release results of oncogenetic report.
5. Patient (or beneficiary) agrees to communicate the contact details of his relatives and that they may be contacted by mail to participate in the LUCID study.
6. Patient affiliated to a Social Health Insurance in France.
7. Patient able to participate and willing to give informed consent prior performance of any study-related procedures.

Exclusion Criteria:

1. No history of hemopathy or no current hemopathy.
2. Patient (or beneficiary) unable to complete questionnaire for social or psychological reasons.
3. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Related cases (Family member):

Inclusion Criteria:

1. Women or man aged ≥ 18 years old.
2. Related to an index case included in the LUCID study.
3. Agreeing to carry out a scientific salivary test for the constitutional research of the DDX41 mutation.
4. Patient affiliated to a Social Health Insurance in France.
5. Patient able to participate and willing to give informed consent prior performance of any study-related procedures.

Exclusion Criteria:

1. Not applicable from version 2 of the protocol. Related in the 4th or 5th degree to an index case included in the LUCID study.
2. Person already identified as an index case in the LUCID study.
3. Person unable to complete questionnaire for social or psychological reasons.
4. Person who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The time to onset of hemopathy defined as the time between the date of birth and the date of diagnosis of an hemopathy. | 74 months after the study start date

SECONDARY OUTCOMES:
Post-transplant relapse-free survival defined as the time between the date of transplantation and the date of all-cause relapse or death. | 74 months after the study start date

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Chu de Bordeaux, Bordeaux
  - Chu de Limoges, Limoges
  - Institut Paoli-Calmettes, Marseille
  - Chu de Montpellier, Montpellier
  - IUCT-O, Toulouse